CLINICAL TRIAL: NCT01058642
Title: A Phase 2A, Randomized, Blinded, Placebo- and Active-controlled, 2-Period Crossover Study to Assess the Analgesic Efficacy, Safety, and Tolerability of ADL5747 in Subjects With Postherpetic Neuralgia
Brief Title: Study to Assess the Efficacy, Safety, and Tolerability of ADL5747 in Participants With Postherpetic Neuralgia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 40CL234
Record Dates: First submitted 2010-01-27; First posted 2010-01-29 (Estimated); Results first posted 2015-07-08 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2015-07

CONDITIONS: Postherpetic Neuralgia
Keywords: pain; delta opioid receptor agonist
MeSH Terms: conditions — Neuralgia, Postherpetic; Pain | interventions — N,N-diethyl-3-hydroxy-4-(spiro(chromene-2,4'-piperidine)-4-yl)benzamide; Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- ADL5747 (Experimental): ADL5747 150 milligrams (mg) administered orally as 1 ADL5747 150-mg capsule and 1 placebo capsule twice daily (BID) for 14 days during 1 of 2 Treatment Periods.
  Interventions: Drug: ADL5747; Drug: Placebo
- Placebo (Placebo Comparator): Placebo: two placebo capsules administered orally BID for 14 days during 1 of 2 Treatment Periods.
  Participants were also administered placebo orally BID during a 14-day washout period that took place between Treatment Period 1 and Treatment Period 2.
  Interventions: Drug: Placebo
- Pregabalin (Active Comparator): Pregabalin administered orally as a dose of 1 pregabalin 75-mg capsule and 1 placebo capsule BID for the first 3 days, increased to a dose of 1 pregabalin 150-mg capsule and 1 placebo capsule BID for the last 11 days of 1 of 2 fourteen-day Treatment Periods, followed by a dose of 1 pregabalin 75-mg capsule and 1 placebo capsule BID for 3 days as a taper period.
  Interventions: Drug: Placebo; Drug: Pregabalin

INTERVENTIONS:
Drug: ADL5747
  Arms: ADL5747
Drug: Placebo
Drug: Pregabalin
  Other Names: Lyrica
  Arms: Pregabalin

SUMMARY:
The primary purpose of this study is to evaluate the analgesic efficacy of ADL5747 in participants with postherpetic neuralgia (PHN). The secondary objective of this study is to evaluate the safety, tolerability, and pharmacokinetics of ADL5747.

ELIGIBILITY:
Key inclusion Criteria:

* have a diagnosis of PHN (defined as pain present for at least 3 months after the healing of herpes zoster rash; there is no upper limit on the duration of PHN)
* have an average daily pain score of at least 4 on the numeric pain rating scale (0-10) at the start of baseline week for Treatment Period 1 (Day -7) through the start of the first week of Treatment Period 1 (Day 1)
* be willing and able to understand and comply with protocol requirements, dietary and dosing regimens, and other protocol instructions and restrictions (for example, forgo use of their normal pain medication and other protocol specified prohibited medications for the duration of the study)
* for male participants, be surgically sterile or agree to use an appropriate method of contraception or have a sexual partner who is surgically sterile or using an insertable, injectable, transdermal, or combination oral contraceptive approved and deemed highly effective by the United States Food and Drug Administration (FDA) from the first dose of study medication through 30 days after the last dose of study medication on Day 49
* for female participants of childbearing potential, be using an insertable, injectable, transdermal, or combination oral contraceptive approved and deemed highly effective by the FDA from the first dose of study medication through 30 days after the last dose of study medication on Day 49 and have negative results on a serum pregnancy test during the start of the screening period to obtain informed consent and determine eligibility for the study (Day -37 to -14) and on a urine pregnancy test during the start of the first week of Treatment Period 1 (Day 1) (women who are surgically sterile [for example, hysterectomy, tubal ligation] or postmenopausal [if ≥ 55 years old, no menses for at least 2 years; if < 55 years old, follicle stimulating hormone concentrations within the postmenopausal range of > 40 milli-International Units per milliliter (mIU/mL) and 17 β estradiol levels of < 37 picograms per milliliter (pg/mL)] are also eligible to participate)

Key Exclusion Criteria:

* be pregnant or lactating
* have significant skin lesions that could interfere with pain assessment
* have a history of seizures or a history of abnormal electroencephalographic results at any time (participants with a history of febrile seizures before the age of 6 years may be enrolled)
* have had previous neurolytic or neurosurgical therapy for PHN
* have had a treatment that included local anesthetic nerve blocks within 30 days before the start of the baseline week for Treatment Period 1 (Day -7)
* have any other type of pain that may impair the self-assessment of pain due to PHN
* have, as determined by the investigator or the sponsor's medical monitor, a history or clinical manifestations of significant renal, hepatic, hematologic, cardiovascular, metabolic, gastrointestinal, neurologic, psychiatric, or other condition that would preclude participation in the study
* have an active malignancy of any type (participants with a history of successfully treated malignancy > 5 years before the scheduled first dose of study medication and participants with treated basal or squamous cell cancer may be enrolled)
* have a medical history or condition that may interfere with drug absorption (for example, stomach resection)
* be currently using protocol specified prohibited medications in the absence of appropriate washout
* be currently taking moderate or strong inhibitors or inducers of cytochrome P450-3A (CYP3A) or inhibitors of P glycoprotein transporters
* have an estimated glomerular filtration rate (GFR) that is less than or equal to 60 mL/min calculated by the Cockcroft Gault equation or have alanine aminotransferase and/or aspartate aminotransferase levels that are at least 2 times the upper limit of normal
* have a history of substance abuse or dependence within the previous 5 years, including alcohol or positive results on the urine drug screen at start of screening period, start of baseline week, or start of the first week of Treatment Period 1 (Day -37 to Day 1); participants may be enrolled if positive results are due to medication(s) prescribed for the participant and permitted by the protocol
* have a history of suicide attempts or be judged clinically to be at serious risk of suicide
* have a score of more than 29 on the Beck Depression Inventory-II at start of screening period (Day -37 to Day -14)
* have a history of allergy to acetaminophen (the rescue medication for this study)
* have a history of intolerance to pregabalin or documented failure to respond to a maximally tolerated dose of pregabalin
* have ever received the investigational drug ADL5747 or have participated in any clinical study involving an investigational product in which they received that product within 30 days before the scheduled administration of study medication for this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2010-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wei Du, MD, Study Director — Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA)
Locations (1):
- Laszlo J. Mate, MD, West Palm Beach, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Sequence 1: Placebo Then Pregabalin: Placebo was administered orally twice daily (BID) to participants for 14 days during Treatment Period 1.
  A two week washout period took place between Treatment Period 1 and Treatment Period 2 where participants were administered placebo orally BID.
  Pregabalin 75 mg BID was administered as 1 pregabalin 75-mg capsule and 1 placebo capsule BID for the first 3 days of Treatment Period 2; the dose was increased to 150 mg BID for the last 11 days of the 2-week treatment period (1 pregabalin 150-mg capsule and 1 placebo capsule BID). This was followed by a dose of pregabalin 75 mg BID (1 pregabalin 75-mg capsule and 1 placebo capsule BID) for 3 days as a taper period followed by placebo orally BID during the last 4 days.
- Treatment Sequence 2: Pregabalin Then Placebo: Pregabalin 75 mg BID was administered as 1 pregabalin 75-mg capsule and 1 placebo capsule BID for the first 3 days of Treatment Period 1; the dose was increased to 150 mg BID for the last 11 days of the 2-week treatment period (1 pregabalin 150-mg capsule and 1 placebo capsule BID).
  At the end of Treatment Period 1 and the start of the first week of the 2-week washout period, participants took a tapered pregabalin dose (75 mg BID) during the first 3 days of the week, followed by placebo orally BID during the last 4 days.
  Placebo was administered orally twice daily (BID) to participants for 14 days during Treatment Period 2.
  At the end of Treatment Period 2, participants received placebo orally BID for 7 days for the taper week.
- Treatment Sequence 3: Placebo Then ADL5747: Placebo was administered orally twice daily (BID) to participants for 14 days during Treatment Period 1.
  A two week washout period took place between Treatment Period 1 and Treatment Period 2 where participants were administered placebo orally BID.
  During Treatment Period 2, ADL5747 150 mg was administered as 1 ADL5747 150-mg capsule and 1 placebo capsule BID for 14 days.
  At the end of Treatment Period 2, participants received placebo orally BID for 7 days for the taper week
- Treatment Sequence 4: ADL5747 Then Placebo: During Treatment Period 1, ADL5747 150 mg was administered as 1 ADL5747 150-mg capsule and 1 placebo capsule BID for 14 days.
  A two week washout period took place between Treatment Period 1 and Treatment Period 2 where participants were administered placebo orally BID.
  Placebo was administered orally twice daily (BID) to participants for 14 days during Treatment Period 2.
  At the end of Treatment Period 2, participants received placebo orally BID for 7 days for the taper week.
Period: Treatment Period 1
Arm/Group | Treatment Sequence 1: Placebo Then Pregabalin | Treatment Sequence 2: Pregabalin Then Placebo | Treatment Sequence 3: Placebo Then ADL5747 | Treatment Sequence 4: ADL5747 Then Placebo
Started | 9 | 12 | 11 | 9
Received at Least 1 Dose of Study Drug | 9 | 12 | 11 | 9
Completed | 7 | 11 | 9 | 7
Not Completed | 2 | 1 | 2 | 2
Not completed — Adverse Event | 0 | 1 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 1
Not completed — Lack of Compliance with Study Drug | 1 | 0 | 0 | 0
Period: Washout Period
Arm/Group | Treatment Sequence 1: Placebo Then Pregabalin | Treatment Sequence 2: Pregabalin Then Placebo | Treatment Sequence 3: Placebo Then ADL5747 | Treatment Sequence 4: ADL5747 Then Placebo
Started | 7 | 11 | 9 | 7
Completed | 7 | 11 | 9 | 7
Not Completed | 0 | 0 | 0 | 0
Period: Treatment Period 2
Arm/Group | Treatment Sequence 1: Placebo Then Pregabalin | Treatment Sequence 2: Pregabalin Then Placebo | Treatment Sequence 3: Placebo Then ADL5747 | Treatment Sequence 4: ADL5747 Then Placebo
Started | 7 | 11 | 9 | 7
Received at Least 1 Dose of Study Drug | 7 | 11 | 9 | 7
Completed | 7 | 11 | 9 | 7
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Treatment Sequence 1: Placebo Then Pregabalin: Placebo: two placebo capsules administered orally BID for 14 days during 1 of 2 Treatment Periods.
  Participants were also administered placebo orally BID during a 14-day washout period that took place between Treatment Period 1 and Treatment Period 2.
  Pregabalin: administered orally as a dose of 1 pregabalin 75-mg capsule and 1 placebo capsule BID for the first 3 days, increased to a dose of 1 pregabalin 150-mg capsule and 1 placebo capsule BID for the last 11 days of 1 of 2 fourteen-day Treatment Periods, followed by a dose of 1 pregabalin 75-mg capsule and 1 placebo capsule BID for 3 days as a taper period.
- Treatment Sequence 2: Pregabalin Then Placebo: Pregabalin: administered orally as a dose of 1 pregabalin 75-mg capsule and 1 placebo capsule BID for the first 3 days, increased to a dose of 1 pregabalin 150-mg capsule and 1 placebo capsule BID for the last 11 days of 1 of 2 fourteen-day Treatment Periods, followed by a dose of 1 pregabalin 75-mg capsule and 1 placebo capsule BID for 3 days as a taper period.
  Placebo: two placebo capsules administered orally BID for 14 days during 1 of 2 Treatment Periods.
  Participants were also administered placebo orally BID during a 14-day washout period that took place between Treatment Period 1 and Treatment Period 2.
- Treatment Sequence 3: Placebo Then ADL5747: Placebo: two placebo capsules administered orally BID for 14 days during 1 of 2 Treatment Periods.
  Participants were also administered placebo orally BID during a 14-day washout period that took place between Treatment Period 1 and Treatment Period 2.
  ADL5747: 150 mg BID administered orally as 1 ADL5747 150-mg capsule and 1 placebo capsule twice daily (BID) for 14 days during 1 of 2 Treatment Periods.
- Treatment Sequence 4: ADL5747 Then Placebo: ADL5747: 150 mg BID administered orally as 1 ADL5747 150-mg capsule and 1 placebo capsule BID for 14 days during 1 of 2 Treatment Periods.
  Placebo: Two placebo capsules administered orally BID for 14 days during 1 of 2 Treatment Periods.
  Participants were also administered placebo orally BID during a 14-day washout period that took place between Treatment Period 1 and Treatment Period 2.
- Total: Total of all reporting groups
Arm/Group | Treatment Sequence 1: Placebo Then Pregabalin | Treatment Sequence 2: Pregabalin Then Placebo | Treatment Sequence 3: Placebo Then ADL5747 | Treatment Sequence 4: ADL5747 Then Placebo | Total
Number analyzed (Participants) | 9 | 12 | 11 | 9 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.8 (8.17) | 58.9 (16.01) | 67.1 (6.98) | 67.4 (8.03) | 62.5 (11.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 7 | 4 | 22
  Male | 2 | 8 | 4 | 5 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 2 | 0 | 2 | 8
  White | 5 | 10 | 11 | 7 | 33
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 12 | 11 | 9 | 41

OUTCOME MEASURES:

1. Primary Outcome: Change in Weekly Average Numeric Pain Rating Scale (NPRS) Score From Baseline to End of Treatment (Week 2 of Each Treatment Period)
Description: The NPRS is an 11-point scale (0 to 10) with 0 indicating no pain and 10 indicating the worst possible pain. The mean of the daily average scores were calculated from the NPRS pain assessments obtained up to 3 times per day over a 7-day period.
Time Frame: Baseline, Week 2 of Treatment Period 1 or 2
Population: Zero participants were analyzed, and no data was collected for this measure. Due to lack of efficacy of ADL5747, the study was terminated early.
Groups:
- ADL5747: ADL5747: 150 milligrams (mg) twice daily administered orally as 1 ADL5747 150-mg capsule and 1 placebo capsule twice daily (BID) for 14 days during 1 of 2 Treatment Periods.
- Placebo: Two placebo capsules administered orally BID for 14 days during 1 of 2 Treatment Periods.
  Participants were also administered placebo orally BID during a 14-day washout period that took place between Treatment Period 1 and Treatment Period 2.
- Pregabalin: Pregabalin: administered orally as a dose of 1 pregabalin 75-mg capsule and 1 placebo capsule BID for the first 3 days, increased to a dose of 1 pregabalin 150-mg capsule and 1 placebo capsule BID for the last 11 days of 1 of 2 fourteen-day Treatment Periods, followed by a dose of 1 pregabalin 75-mg capsule and 1 placebo capsule BID for 3 days as a taper period.
Arm/Group | ADL5747 | Placebo | Pregabalin
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Description: Adverse events are summarized by study drug for participants who received at least 1 dose of that study drug. For example, 9 participants from Treatment Sequence (TS) 4 received at least 1 dose of ADL5747 in Treatment Period (TP) 1, and 9 participants from TS 3 received at least 1 dose ADL5747 in TP 2. Therefore, 18 participants received ADL5747.
Arm/Group | ADL5747 | Placebo | Pregabalin
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/38 | 0/19
Other Adverse Events (participants affected / at risk) | 4/18 | 7/38 | 9/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ADL5747 (N=18) | Placebo (N=38) | Pregabalin (N=19)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 5 (5)
Dry Mouth (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Gait Disturbance (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1)
Somnolence (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (3)
Euphoric mood (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Fatigue (General disorders) | 1 (1) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dysarthria (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Edema peripheral (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Feeling jittery (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoesthesia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoesthesia oral (General disorders) | 0 (0) | 1 (1) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nystagmus (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Paresthesia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Speech disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Urine analysis abnormal (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
On the basis of the interim analysis, the results indicated that ADL5747 did not show sufficient efficacy to continue the study; therefore, formal and final efficacy analyses were not generated for this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other